CLINICAL TRIAL: NCT00738231
Title: Two Distinct Training Methods for Healthy Heart in Low Social and Economical Society
Brief Title: Training Methods for a Doctrine Of Life With Healthy Heart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Selma Metintas, MD, PhD, ESOGU
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2007/37
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Last update posted 2009-06-19 (Estimated); Status verified 2008-08

CONDITIONS: Heart Diseases
Keywords: risk factors; coronary arterial hearth disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): Group I's training material consisted of a brochure with the information we wanted the public to know about heart disease. The brochure had such titles as "Cardiovascular Diseases, let us protect our hearts, the importance of cholesterol in preventing heart diseases, watch out for blood pressure, quit smoking for your health, weight watching, nutrition, food to avoid in cardiovascular disease, an easy method: exercise and exercise control, and an appropriate body weight vs. height chart for adults"
  Interventions: Behavioral: Training
- II (Active Comparator): The Group II training material document was a letter in the form of a prescription in which the individual was addressed by name, the risk factors established at the first stage were explained, and the suggested measures for protection from such risk factors were indicated.
  Interventions: Behavioral: Training

INTERVENTIONS:
Behavioral: Training — The training materials were randomly distributed to study participant groups. The list of names was systematically divided into two groups: odd-numbered individuals were given brochures only, and even-numbered individuals were given both letters and brochures. Since we could not have prevented an illustrated material to be passed by in a closed environment, it was deemed appropriate to distribute both the letter and brochure instead of just the brochure.
  Other Names: CAHD; TM
  Arms: I
Behavioral: Training — The training materials were randomly distributed to study participant groups. The list of names was systematically divided into two groups: odd-numbered individuals were given brochures only, and even-numbered individuals were given both letters and brochures. Since we could not have prevented an illustrated material to be passed by in a closed environment, it was deemed appropriate to distribute both the letter and brochure instead of just the brochure.
  Other Names: CAHD; TM
  Arms: II

SUMMARY:
This study is an interventional study which was conducted in the field. The investigators intended to develop an efficient and economically valuable method which can decrease the risk factors for prevention of cardiovascular diseases. Effective control of cardiovascular diseases necessitates a salutogenetic approach to develop efficient and cheap methods to decrease risk factors.

In this study, the aim of preparing the Group II training material was to enable the individual to see his or her risks as unique, and to proceed with life by adapting personal behaviors. Group II's training material was formatted as a prescription. Because giving a prescription for a doctor is very important in low socioeconomical group person.

This study showed that social programs oriented towards individual behavioral changes assume an important role in decreasing cardiovascular risk factors.

DETAILED DESCRIPTION:
Background:

Effective control of cardiovascular diseases necessitates a salutogenetic approach to develop efficient and economical methods to decrease risk factors.

Methods:

This study was conducted in three stages in a semi-rural region of Eskisehir, Turkey. In the first stage, individuals selected by random sampling were evaluated in terms of social-demographic characteristics and the risk factors present for cardiovascular diseases. A scale comprised of 19 questions was implemented for data assessment. In the second stage, training materials were randomly distributed. Group I's training material consisted of a brochure containing pictures and general information on heart disease; Group II members additionally received a personalized letter that further explained their individual risk factors and suggested measures for increased protection and prevention - in short, Group II's training material was formatted as a prescription. In the third stage, the subjects were screen against the cardiovascular risks factors one year later to assess and determine if there had been any changes in their attitudes towards the dangers of the cardiovascular diseases.

ELIGIBILITY:
Inclusion Criteria:

* Over 40 years of age were contacted.
* Individuals who were literate or had at least one literate person in the household were selected through random sampling via the records of local health care units.

Exclusion Criteria:

* Under 40 years of age and immigrants

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Increase of score of the knowledge about the risk factors for cardiovascular diseases | 1 month

SECONDARY OUTCOMES:
Stop smoking; to regulate of arterial tension; properly change of feeding behaviour | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Selma Metintas, MD,Prof., Study Chair — ESOGU
Locations (1):
- ESOGU, Eskişehir, Turkey (Türkiye)

REFERENCES:
- See also: Eskisehir Osmangazi University — http://www.ogu.edu.tr/